CLINICAL TRIAL: NCT01290536
Title: Safety Profile Assessment of TheraSphere® Yttrium-90 Glass Microspheres Used for Treatment of Metastatic Liver Disease From Primary Colorectal, Neuroendocrine, Cholangiocarcinoma, Melanoma, and Breast Cancers Refractory to Chemotherapy: A Pilot Study
Brief Title: Yttrium-90 Radioembolization Using Glass Microspheres (TheraSphere) for Patients With Liver Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nicholas Fidelman, MD (Other)
Responsible Party: Sponsor-Investigator, Nicholas Fidelman, MD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSF-SIRT-Metastases
Record Dates: First submitted 2011-02-01; First posted 2011-02-07 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Neoplasms; Neuroendocrine Tumors; Cholangiocarcinoma; Melanoma; Breast Cancer
Keywords: Liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neuroendocrine Tumors; Cholangiocarcinoma; Melanoma; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Yttrium-90 liver radioembolization (Experimental)
  Interventions: Device: Selective internal radiation therapy to the liver using Yttrium-90 glass microspheres (TheraSphere)

INTERVENTIONS:
Device: Selective internal radiation therapy to the liver using Yttrium-90 glass microspheres (TheraSphere) — Administration of Yttrium-90 glass microspheres (TheraSphere) into the hepatic artery

SUMMARY:
This is a prospective pilot study designed to document safety and efficacy of liver-directed therapy for colorectal, neuroendocrine, cholangiocarcinoma, melanoma, and breast cancer metastases to the liver using Yttrium-90 glass microspheres (TheraSphere).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic colorectal, neuroendocrine, cholangiocarcinoma, melanoma, or breast malignancy with liver dominant disease. Diagnosis may be made by histo- or cyto-pathology, or by clinical and imaging criteria.
* The cancer is unresectable.
* All patients must be off all chemotherapeutic regimens for 30 days prior to and 30 days after TheraSphere treatment. Concurrent therapy with octreotide is permitted, when appropriate.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Age 18 years or older.
* Able to understand informed consent.

Exclusion Criteria:

* Evidence of potential delivery of greater than 16.5 mCi (30 Gy absorbed dose) of radiation to the lungs on either:

  * single TheraSphere administration; or
  * cumulative delivery of radiation to the lungs greater than 50 Gy over multiple treatments.
* Evidence of any detectable Tc-99m macroaggregated albumin deposition in the stomach or duodenum, after application of established angiographic techniques to stop such deposition.
* Previous radiation therapy to the lungs and/or to the upper abdomen
* Pregnancy
* Symptomatic lung disease.
* Significant extrahepatic disease representing an imminent life-threatening outcome.
* Active uncontrolled infection
* Any pre-treatment laboratory findings within 30 days of treatment demonstrating:

  * Aspartate or alanine aminotransferase level greater than 5 times upper normal limit.
  * Serum bilirubin greater than 2 mg/dl
  * Infiltrative tumor on imaging
  * Tumor volume greater than 70% of liver volume
  * Tumor volume greater than 50% of liver volume and serum albumin level less than 3 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 2010 and October 2013, 42 adult patients with liver-dominant metastaticd colorectal or neuroendocrine cancer to the liver, or intrahepatic cholangiocarcinoma were enrolled in a prospective single-institution pilot study.
Groups:
- Yttrium-90 Radioembolization: Selective internal radiation therapy using Yttrium-90 glass microspheres (TheraSphere)
Period: Overall Study
Arm/Group | Yttrium-90 Radioembolization
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: per protocol
Arm/Group | Yttrium-90 Radioembolization
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] | 61 [35 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse effects of treatment with Yttrium-90 glass microspheres (TheraSphere) were collected prospectively for 6 months after each treatment administration.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Yttrium-90 Radioembolization
Number analyzed (Participants) | 42
participants | 42

2. Secondary Outcome: Radiographic Response
Description: Radiographic response of treated lesions on cross-sectional imaging (computed tomography or magnetic resonance imaging) following treatment with Yttrium-90 glass microspheres (TheraSphere) was assessed based on Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no change in target lesions; Progressive Disease (PD), increase in target lesions.
Time Frame: 6 months after treatment
Population: Response data are presented by primary disease sites: Colorectal (mCRC), Neuroendocrine (NET), and all other tumors. One patient with mCRC did not have follow-up cross-sectional imaging. Therefore, radiographic response data was available for 20 of 21 patients with mCRC.
Measure: Number; unit: participants
Groups:
- Colorectal - Yttrium-90 Radioembolization; Neuroendocrine - Yttrium-90 Radioembolization; Other Tumors - Yttrium-90 Radioembolization: Selective internal radiation therapy using Yttrium-90 glass microspheres (TheraSphere)
Arm/Group | Colorectal - Yttrium-90 Radioembolization | Neuroendocrine - Yttrium-90 Radioembolization | Other Tumors - Yttrium-90 Radioembolization
Number analyzed (Participants) | 20 | 11 | 10
participants
  Complete Response (CR) | 0 | 0 | 0
  Partial Response (PR) | 4 | 7 | 1
  Stable Disease (SD) | 12 | 4 | 6
  Progressive Disease (PD) | 4 | 0 | 3

ADVERSE EVENTS:
Time Frame: 6 months after treatment
Groups:
- Yttrium-90 Liver Radioembolization: Selective internal radiation therapy using Yttrium-90 glass microspheres (TheraSphere)
Arm/Group | Yttrium-90 Liver Radioembolization
Serious Adverse Events (participants affected / at risk) | 3/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Yttrium-90 Liver Radioembolization (N=42)
hospitalization for carcinoid crisis (Blood and lymphatic system disorders) | 1/11 (1) — Only patients with neuroendocrine tumors were at risk for carcinoid crisis. Therefore denominator for this adverse event is 11, not 42.
Vomiting (Gastrointestinal disorders) | 1 (1) — grade 3
gastric ulcer (Gastrointestinal disorders) | 1 (1) — grade 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Yttrium-90 Liver Radioembolization (N=42)
Lymphopenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Arrhythmia (Cardiac disorders) | 1
PT/INR (Blood and lymphatic system disorders) | 1 — Coagulation
Fatigue (General disorders) | 34
Fever (General disorders) | 6
Rigors (General disorders) | 1
Sweating (General disorders) | 7
Flushing (General disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Anorexia (Gastrointestinal disorders) | 18
Diarrhea (Gastrointestinal disorders) | 3
Nausea (General disorders) | 20
Ulcer (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 8
Edema (Blood and lymphatic system disorders) | 1
Albuminemia (Metabolism and nutrition disorders) | 15
ALT (Metabolism and nutrition disorders) | 14
AST (Metabolism and nutrition disorders) | 24
Bilirubin (Metabolism and nutrition disorders) | 9
Creatinine (Metabolism and nutrition disorders) | 4
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Abdominal pain (General disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No